CLINICAL TRIAL: NCT06201156
Title: Comparison of Pulmonary Index Score After Treatment With Salbutamol Through Nebulizers vs Metered-Dose Inhalers With Spacer Device For Treatment Of Childhood Wheeze
Brief Title: Comparison of Nebulizers vs Metered-Dose Inhalers With Spacer Device For Treatment Of Childhood Wheeze
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Arooj Khan, Post Graduate Resident, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 847/DME/KMC
Record Dates: First submitted 2023-12-15; First posted 2024-01-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Childhood Asthma With Acute Exacerbation
MeSH Terms: interventions — Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A / Nebulizer Group (Active Comparator): Group A/ Nebulizer group will receive 3 puffs of a placebo MDI with a spacer, followed immediately by a standard dose of 0.15 mg/kg of salbutamol in 3 mL of isotonic sodium chloride solution delivered by an oxygen-driven nebulizer at a flow rate of 6 L/min.
  Interventions: Device: Metered Dose Inhaler With Spacer Device
- Group B / MDI with Spacer Device Group (Experimental): Group B/ MDI with Spacer Group will receive 3 puffs (90 pg per puff) of salbutamol MDI with a spacer, followed by 3 mL of nebulized isotonic sodium chloride solution. All treatments will be given at 20-minute intervals.
  Interventions: Device: Metered Dose Inhaler With Spacer Device

INTERVENTIONS:
Device: Metered Dose Inhaler With Spacer Device — Bronchodilator Therapy

SUMMARY:
The goal of this randomized controlled trial is to compare two different devices for the administration of the standard protocol drug. The main question it aims to answer is are metered dose inhalers with spacer device as effective as nebulization with salbutamol in treatment of childhood wheeze

Children will be divided in two groups using block randomization method. Children in group A will be nebulizer group, treatment will consist of 3 puffs of a placebo MDI with a spacer, followed immediately by a standard dose of 0.15 mg/kg of salbutamol in 3 mL of isotonic sodium chloride solution delivered by an oxygen-driven nebulizer at a flow rate of 6 L/min.

For patients in group B spacer group, treatment consisted of 3 puffs (90 pg per puff) of salbutamol MDI with a spacer, followed by 3 mL of nebulized isotonic sodium chloride solution. All treatments will be given at 20-minute intervals. For administration of the MDI, the investigator will dispense I puff of salbutamol or placebo into the spacer and held the mask on the child's face while the child breathed 5 to 6 times through the mask. This process will b-e repeated for a total of 3 puffs per treatment. All patients will be treated by the principal investigator, at end of treatment need for admission and pulmonary index will be noted.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 6 to 24 months

* Patients of both gender
* Patients presenting to emergency department with bilateral wheeze

Exclusion Criteria:

Patients with history of chronic lung condition (including congenital anomalies, cystic fibrosis, and bronchopulmonary dysplasia).

* Patients with history of congenital heart disease.
* Patients with history of intubation for longer than 1 week during the neonatal period.
* Patients having symptoms consistent with croup.
* Patients with signs of impending respiratory failure i.e Pulmonary index score of 12.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
compare mean pulmonary index score after treatment with salbutamol through nebulizers vs metered dose inhalers | 1 hour
  primary outcome is defined as Comparison of mean pulmonary index score after treatment with salbutamol through nebulizers vs metered dose inhalers with spacers for treatment of wheezing in children aged 6 to 24 months in a pediatric emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Arooj Khan, MBBS, Principal Investigator — Khyber Teaching Hospital
Locations (1):
- Khyber Teaching Hospital, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 months

REFERENCES:
- [Background] Csonka P, Tapiainen T, Makela MJ, Lehtimaki L. Optimal administration of bronchodilators with valved holding chambers in preschool children: a review of literature. Eur J Pediatr. 2021 Oct;180(10):3101-3109. doi: 10.1007/s00431-021-04074-3. Epub 2021 Apr 20. PMID 33877400
- [Background] Nurmagambetov T, Kuwahara R, Garbe P. The Economic Burden of Asthma in the United States, 2008-2013. Ann Am Thorac Soc. 2018 Mar;15(3):348-356. doi: 10.1513/AnnalsATS.201703-259OC. PMID 29323930
- [Background] Roncada C, Andrade J, Bischoff LC, Pitrez PM. COMPARISON OF TWO INHALATIONAL TECHNIQUES FOR BRONCHODILATOR ADMINISTRATION IN CHILDREN AND ADOLESCENTS WITH ACUTE ASTHMA CRISIS: A META-ANALYSIS. Rev Paul Pediatr. 2018 Jul-Sep;36(3):364-371. doi: 10.1590/1984-0462/;2018;36;3;00002. Epub 2018 Jul 10. PMID 29995144
- [Background] Alharbi AS, Yousef AA, Alharbi SA, Al-Shamrani A, Alqwaiee MM, Almeziny M, Said YS, Alshehri SA, Alotaibi FN, Mosalli R, Alawam KA, Alsaadi MM. Application of aerosol therapy in respiratory diseases in children: A Saudi expert consensus. Ann Thorac Med. 2021 Apr-Jun;16(2):188-218. doi: 10.4103/atm.atm_74_21. Epub 2021 Apr 17. PMID 34012486
- [Background] Payares-Salamanca L, Contreras-Arrieta S, Florez-Garcia V, Barrios-Sanjuanelo A, Stand-Nino I, Rodriguez-Martinez CE. Metered-dose inhalers versus nebulization for the delivery of albuterol for acute exacerbations of wheezing or asthma in children: A systematic review with meta-analysis. Pediatr Pulmonol. 2020 Dec;55(12):3268-3278. doi: 10.1002/ppul.25077. Epub 2020 Sep 25. PMID 32940961
- [Background] Schell DN, Durham D, Murphree SS, Muntz KH, Shaul PW. Ontogeny of beta-adrenergic receptors in pulmonary arterial smooth muscle, bronchial smooth muscle, and alveolar lining cells in the rat. Am J Respir Cell Mol Biol. 1992 Sep;7(3):317-24. doi: 10.1165/ajrcmb/7.3.317. PMID 1325812
- [Background] Dimino, K. Using A Metered Dose Inhaler (Mdi) With Spacer or Nebulizer for Managing Children Under 5 Years of Age with Exacerbation of Wheezing or Asthma. 2019; 11(2): 555815.10.19080/JOJNHC.2019.11.555815